CLINICAL TRIAL: NCT02901470
Title: Observational Study of the Incidence of Pressure Ulcers on the Help Support of Prevention of Bedsores POLYAIR®
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2015/EV-02
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The support of help to the prevention of sores include a big diversity of devices. The clinical experiment of these support comes up against the problem of the large number of factors participants in the genesis of bedsores. Nevertheless, it seems to be interesting to estimate the incidence of bedsores in these supports, with control of other factors

ELIGIBILITY:
Inclusion Criteria:

* Norton Index <9,
* No sores in ischiatic zone,
* Sitting position not less than 2 hours per day

Exclusion Criteria:

* Sores in ischiatic zone,
* Sitting position >2 hours per day

Ages: 20 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who are hospitalized in CHU of Nîmes with high risk of sores (Norton <9)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of sores in ischiatic zone | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nîmes, Nîmes, GARD, France